CLINICAL TRIAL: NCT01739790
Title: Effects of High-Dose N-Acetylcysteine on Respiratory Health Status in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Chronic Bronchitis: A Randomized, Placebo-Controlled Trial-3
Brief Title: N-Acetylcysteine for Patients With COPD and Chronic Bronchitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI discretion
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1210M21542
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: COPD; Chronic Bronchitis
Keywords: COPD; Chronic Bronchitis; N-acetylcysteine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): Identical placebo pills twice daily for 8 weeks Placebo pills manufactured to mimic appearance of intervention drug n-acetylcysteine and prescribed with identical frequency and duration.
  Interventions: Drug: Placebo
- N-Acetylcysteine (Active Comparator): 1800 mg twice daily for 8 weeks
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — 1800 mg twice daily for 8 weeks
  Arms: N-Acetylcysteine
Drug: Placebo — Identical placebo manufactured to mimic appearance of intervention drug with identical frequency and duration.
  Arms: Sugar Pill

SUMMARY:
N-acetylcysteine (NAC) is described as having mucolytic and antioxidant properties. It is widely prescribed for patients with chronic obstructive lung disease (COPD), particularly for those who have accompanying symptoms of chronic cough and sputum production. Compared to placebo, high-dose NAC will improve Saint George Respiratory Questionnaire scores in patients with COPD and chronic bronchitis.

DETAILED DESCRIPTION:
A total of 130 subjects with COPD and chronic bronchitis will be randomized (in a double-blind fashion) to receive either high-dose NAC (1800 mg) or matching placebo twice daily for eight weeks. Respiratory health status, assessed by changes in St. George's Respiratory Questionnaire, will be used to determine the effects of NAC on lung function. It is anticipated that the subjects on high dose NAC will have improved scores.

ELIGIBILITY:
Inclusion Criteria:

* Capability to provide written informed consent
* Age ≥ 40 years and ≤ 85 years
* FEV1/FVC ratio (post bronchodilator) < 70%
* FEV1 (post bronchodilator) < 65%
* Presence of chronic cough and sputum production defined as the following:
* Presence of chronic cough and sputum will be defined by responses to the first two questions on the SGRQ. Subjects who respond positively to both question 1 (cough) and question 2 (sputum) on the SGRQ as either "several days per week" or "almost every day" will be eligible
* Current or former smoker with lifetime cigarette consumption of at least 10 pack-years
* Negative serum pregnancy test at the baseline visit if patient is a pre-menopausal female (menopause defined as absence of a menstrual cycle in the last 12 months)
* Must be fluent in speaking the English language

Exclusion Criteria:

* Not fully recovered for at least 30 days from a COPD exacerbation characterized by typical symptoms and treated with antibiotics or prednisone
* Known allergy or sensitivity to NAC or albuterol
* Any patient with unstable cardiac disease
* Any patient with a documented history of uncompensated congestive heart failure in the last 2 years
* Clinical diagnosis of asthma, bronchiectasis, cystic fibrosis, or severe alpha-1 antitrypsin deficiency
* Active lung cancer or history of lung cancer if it has been less than 2 years since lung resection or other treatment. If history of lung cancer, must have no evidence of recurrence in the 2 years preceding the baseline visit.
* Undergoing active treatment for malignancy except for hormonal therapy (i.e. prostate cancer, breast cancer) or non-metastatic skin cancer and are not symptomatic
* Chronic kidney disease with an estimated GFR of < 30 ml/min. GFR will be estimated using the Modification of Diet in Renal Disease (MDRD) formula
* History of cirrhosis with evidence of portal hypertension (ascites, chronic edema)
* Participation in a pulmonary rehabilitation program or completion within past 6 weeks
* Prisoners or institutionalized patients
* Participation in another study involving an investigational product within 30 days of the baseline visit
* Pregnant or breast-feeding patients.
* Use of guaifenesin in the last 30 days
* Currently on long acting nitrates for angina or heart failure
* Abnormalities in screening blood work defined as:
* WBC < 3.0 or > 15.0 K/cmm
* Hemoglobin < 9.0 or > 17.0 gm/dl
* Platelets < 75 or > 400 K/cmm
* ALT > 3 times the upper limit of normal
* INR > 1.5 unless on warfarin therapy
* Any concomitant condition that might endanger the patient through participation in the study or interfere with study procedures, as assessed by the investigator

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis E Niewoehner, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johnson K, McEvoy CE, Naqvi S, Wendt C, Reilkoff RA, Kunisaki KM, Wetherbee EE, Nelson D, Tirouvanziam R, Niewoehner DE. High-dose oral N-acetylcysteine fails to improve respiratory health status in patients with chronic obstructive pulmonary disease and chronic bronchitis: a randomized, placebo-controlled trial. Int J Chron Obstruct Pulmon Dis. 2016 Apr 21;11:799-807. doi: 10.2147/COPD.S102375. eCollection 2016. PMID 27143871

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | N-Acetylcysteine
Started | 24 | 27
Completed | 22 | 23
Not Completed | 2 | 4
Not completed — Early Trial Termination | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | N-Acetylcysteine | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Continuous [Mean (Full Range); unit: Years] | 68.9 [60.7 to 77.1] | 70.1 [62.4 to 77.8] | 69.5 [60.7 to 77.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Saint George's Respiratory Questionnaire
Description: The St. George's Respiratory Questionnaire (SGRQ) is scored on a scale of 1 to 100 with 100 representing the worst respiratory health status. The instrument is self-administered at baseline and again after 8-weeks of treatment.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | N-Acetylcysteine
Number analyzed (Participants) | 22 | 23
units on a scale
  Change in SGRQ Symptoms | -9.8 (17.8) | -3.5 (18.6)
  Change in SGRQ Activity | -3.7 (14.5) | -4.0 (13.6)
  Change in SGRQ Impact | -7.5 (20.1) | -4.5 (19.9)
  Change in SGRQ Total | -7.1 (16.1) | -3.9 (12.1)
Statistical Analysis 1: Comparison: Placebo vs N-Acetylcysteine; Test type: Other; p = 0.45, Fisher Exact

ADVERSE EVENTS:
Arm/Group | Placebo | N-Acetylcysteine
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23
Serious Adverse Events (participants affected / at risk) | 2/22 | 3/23
Other Adverse Events (participants affected / at risk) | 9/22 | 13/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | N-Acetylcysteine (N=23)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=22) | N-Acetylcysteine (N=23)
Rotator cuff repair (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Alcohol abuse (Social circumstances) | 1 (1) | 0 (0)
Ruptured Baker's cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Worsening Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Increased shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Edema (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Weight Loss (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Face rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Worsening Prostatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral stricture (Renal and urinary disorders) | 0 (0) | 1 (1)
Abdominal pain (General disorders) | 0 (0) | 1 (1) — Post pulmonary function tests
Influenza (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No